CLINICAL TRIAL: NCT03669562
Title: The Safety, Tolerability and Pharmacokinetic Phrase I Study of Alprostadil Fat Emulsiom Injection in Healthy Adult Volunteers
Brief Title: The Safety and Tolerability of Alprostadil Liposome for Injection in Healthy Adult Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLDE201801/PRO
Record Dates: First submitted 2018-08-21; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Lower Extremity Arterial Occlusive Diseases
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alprostadil liposome (Experimental)
  Interventions: Drug: Alprostadil Liposome for Injection
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alprostadil Liposome for Injection — intravenous infusion Alprostadil Liposome
  Arms: Alprostadil liposome
Drug: Placebo — intravenous infusion liposome control
  Arms: Placebo

SUMMARY:
Conducted in Chinese healthy adult volunteers,the study aims to observe the safety, tolerability and pharmacokinetic of single-dose administration of different doses of Alprostadil Liposome for Injection as well as to confirm the safety dose range.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers are at least 18 years of age and no older than 40.
* BMI are at least 19.0kg/m2,and no more than 24.0kg/m2.(The male weight is greater than or equal to 50kg.The female weight is greater than or equal to 50kg.)Subjects who are overweight or underweight will not be inclusion.
* Subjects with normal medical history,vital signs,physical examination and clinical examination (routine blood,routine urine,blood chemistry,coagulation function and ECG,X-ray,intraocular pressure and so on).
* A negative hepatitis B surface antigen,hepatitis C,HIV or syphilis test result.
* Subjects with the ability to communicate with investigators.Besides,subjects must be willing to remain at the study center as required per protocal to complete all visit assessments.

Exclusion Criteria:

* Subjects have brain dysfunction,mental development disorders or speech disorders that unable to communicate with investigators.
* Subjects with a history of psychiatric disease or drug dependence.
* Subjects with a medical history about cardiac,liver,renal,digestive system or neurological.
* Subjects with the family history of diabetes,the history of pancreatitis,cholelithiasis or asthma.
* Subjects significantly abuse alcohol or tobacco.
* Drink in 24 hours before post-dosing of study drug.
* Subjects who had taken medications within 2 weeks.
* Subjects who had suffer from exsanguine or donated blood over 400ml within 3 months will be excluded.
* Subjects who participate in other clinical trials within 3 months will be excluded.
* History of hypersensitivity or allergy to any of the study drugs or to drugs of similar chemical classes.
* Subjects with a history of fainting.
* Subjects who had infected for unknown reason.
* Subjects with interstitial pneumonia.
* Subjects with glaucoma or intraocular pressure with hyperthyroidism.
* Women who are pregnant or lactating.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-08-07 (Actual); Primary Completion 2018-10-15 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 8 days
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Xuhuiqu central hospital, Shanghai, Shanghai Municipality, China